CLINICAL TRIAL: NCT03131115
Title: Lateral Crural Strut Graft vs Bone-Anchored Suspension for Treatment of Lateral Nasal Wall Insufficiency: A Randomized Clinical Trial.
Brief Title: Lateral Crural Strut Graft vs Bone-Anchored Suspension for Treatment of Lateral Nasal Wall Insufficiency
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to enroll patient
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sam P. Most, Division of Facial Plastic and Reconstructive Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 39000
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Nasal Valve Incompetence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lateral Crural Strut Graft (Active Comparator): Lateral crura strut graft is a well described and universally used technique involves strengthening lateral crus of lower lateral cartilage of the nose with piece of cartilage.
  Interventions: Procedure: Lateral Crural Strut Graft
- Bone-Anchored suspension (Active Comparator): Bone- Anchored suspension is a well described surgical technique which involves anchoring the nasal sidewall to the bony rim below the eye.
  Interventions: Procedure: Bone Anchored Suspension

INTERVENTIONS:
Procedure: Lateral Crural Strut Graft — surgical technique as described
  Other Names: LCSG ( lateral crural strut graft)
  Arms: Lateral Crural Strut Graft
Procedure: Bone Anchored Suspension — Surgical technique as described
  Other Names: BAST(Bone Anchored Suspension technique)
  Arms: Bone-Anchored suspension

SUMMARY:
Lateral nasal wall insufficiency is a source of nasal obstruction which plagues many people as the sidewall of the nose collapses due to negative pressure and structural weaknesses of the nose. Bone anchored suture suspension is used by many surgeons to treat it, and involves anchoring the nasal sidewall to the bony rim below the eye. Lateral crura strut graft is another well described and universally used technique involves strengthening lateral crus of lower lateral cartilage of the nose with piece of cartilage. This study aims to compare the two well known and universally used treatments to each other. Based on expert opinions these procedures are both safe and efficient but given lack of randomized clinical trials comparing these 2 techniques, it is difficult to extrapolate which procedure is superior.

DETAILED DESCRIPTION:
Patients with lateral nasal wall collapse who are eligible for surgical repair will be presented with the opportunity to participate. Once consented, standard pre-operative evaluation will be performed including evaluation of degree of lateral nasal wall collapse. They will also be screened with validated quality of life screening tools for nasal congestion, which include the NOSE scale and a visual analog scale. They will then be randomized to treatment either with Lateral crura strut graft or bone anchored suture suspension, in combination with likely other areas of functional rhinoplasty such as septoplasty and turbinate reduction. All of our patients will be seen 1 week, 2-3 month and 1 year after surgery

ELIGIBILITY:
Inclusion Criteria:

- Eligible subjects with be healthy, adults with lateral nasal wall collapse with or without septal deviation, turbinate hypertrophy, or narrowed internal nasal valve. They must have failed prior medical management with topical nasal steroid or topical or oral antihistamines. They must be able to read, sign, and demonstrate understanding of the research protocol, including agreement to randomization for treatment of their lateral nasal wall collapse

Exclusion Criteria:

* All subjects shall be excluded with evidence or history of prior rhinoplasty, immunocompromise, smokers, chronic sinusitis, history of radiation to the head and neck, septal perforation, granulomatous disease, or pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
NOSE (Nasal Obstruction Symptom Evaluation)score change from baseline to 12 months post op | 1 year
  Nasal Obstruction Symptom Evaluation (NOSE) scale is a validated disease-specific questionnaire for the assessment of Nasal Obstruction (NO)

SECONDARY OUTCOMES:
Visual Analogue Scale for nasal obstruction | 1 year
  The scale is a 10-cm horizontal line anchored by word descriptors. It is scored by measuring the distance in millimeters from the left of where the patient's mark was placed. A higher number indicates more severe symptoms.
Visual analogue scale for satisfaction with appearance of the nose | 1 year
  The scale is a 10-cm horizontal line anchored by word descriptors. It is scored by measuring the distance in millimeters from the left of where the patient's mark was placed. A higher number indicates higher degree of satisfaction
physician derived lateral wall insufficiency grading system | 1 year
  This is a validated grading system which is measured by physician based on degrees of nasal valve insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: Sam P Most, MD, Principal Investigator — Stanford University
Locations (1):
- Division of Facial Plastics and Reconstructive Surgery, Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD

REFERENCES:
- [Background] Stewart MG, Witsell DL, Smith TL, Weaver EM, Yueh B, Hannley MT. Development and validation of the Nasal Obstruction Symptom Evaluation (NOSE) scale. Otolaryngol Head Neck Surg. 2004 Feb;130(2):157-63. doi: 10.1016/j.otohns.2003.09.016. PMID 14990910
- [Background] Tsao GJ, Fijalkowski N, Most SP. Validation of a grading system for lateral nasal wall insufficiency. Allergy Rhinol (Providence). 2013 Summer;4(2):e66-8. doi: 10.2500/ar.2013.4.0054. PMID 24124639
- [Background] Most SP. Comparing Methods for Repair of the External Valve: One More Step Toward a Unified View of Lateral Wall Insufficiency. JAMA Facial Plast Surg. 2015 Sep-Oct;17(5):345-6. doi: 10.1001/jamafacial.2015.0790. No abstract available. PMID 26247486